CLINICAL TRIAL: NCT05857579
Title: Diamond Bur Microblepharoexfoliation Combined With Intense Pulse Light and Meibomian Gland Expression for Evaporative Dry Eye: A Short-term Controlled Study
Brief Title: Diamond Bur Microblepharoexfoliation, Intense Pulse Light and Meibomian Gland Expression for Evaporative Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Antonio Ballesteros Sánchez, Principal Investigator, University of Seville
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIVIUS-ABS-001
Record Dates: First submitted 2023-04-08; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Dry Eye Disease
Keywords: Microblepharoexfoliation; Intense pulse light; Meibomian gland expression; Meibomian gland dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MBE-IPL-MGX treatment and home-based therapy. (Experimental): In this arm, participants received three sessions of MBE-IPL-MGX treatment and home-based therapy.
  Interventions: Procedure: Microblepharoexfoliation; Procedure: Intense pulse light; Procedure: Meibomian gland expression; Drug: Home-based therapy
- Home-based therapy (Active Comparator): In this arm, participants received home-based therapy alone.
  Interventions: Drug: Home-based therapy

INTERVENTIONS:
Procedure: Microblepharoexfoliation — MBE was performed using the yokefellow instrument (Youke Electronic Corporation, Guangzhou, China), which contains a handpiece with a 1.80 mm diameter medical-grade diamond bur. Patients underwent MBE on the upper and lower lid margin of both eyes at 500 rpm until complete removal of accumulated biofilm debris, epithelial keratinization or capped meibomian glands. MBE was carried out only in the first combined treatment session.
  Other Names: MBE
  Arms: MBE-IPL-MGX treatment and home-based therapy.
Procedure: Intense pulse light — IPL treatment was carried out with Thermaeye Plus (MDS Medical Technologies SL, Barcelona, Spain). The procedure began by applying an ultrasound gel (Carmado SL, Alicante, Spain) to the patient's periocular areas and upper eyelids. In the periocular areas, 6 light pulses were applied; 4 light pulses on the skin below the lower eyelid (with handpiece placed horizontally in the first pass and vertically in the second pass) and 2 light pulses on the canthal area (with handpiece placed vertically in first and second pass). The parameters were as follows: (1) Filter: 650 nm; (2) fluence: 9 j/cm2; (3) pulses: 2; (4) duration: 3 ms; (5) Delay: 20 ms; and (6) Cooling: 70%. In the upper eyelids, 4 light pulses were applied; 2 light pulses in the first and second pass, respectively. The parameters were as follows: (1) Filter: 650 nm; (2) Fluence: 5 j/cm2; (3) pulses: 1; (4) duration: 3 ms and (5) Cooling: 70%.
  Other Names: IPL
  Arms: MBE-IPL-MGX treatment and home-based therapy.
Procedure: Meibomian gland expression — Finally, the MGX was performed on both upper and lower eyelids of each eye with a Collins forceps (Medi Instrument Inc, New York, USA).
  Other Names: MGX
  Arms: MBE-IPL-MGX treatment and home-based therapy.
Drug: Home-based therapy — Home-based therapy was based on Therapearl eye mask warming compress (Bausch & Lomb, Madrid, Spain) twice a day and Eyestil synfo eyedrops (Sifi Iberica SL, Madrid, Spain) 4 times a day during the study
  Other Names: HBT

SUMMARY:
The goal of this clinical trial is to assess the efficacy and safety of microblepharoeexfoliation (MBE), intense pulse light (IPL) and meibomian gland expression (MGX) combination in patients with meibomian gland dysfunction (MGD).

The main question it aims to answer are:

* Does MBE-IPL-MGX treatment improve dry eye symptoms?
* Does MBE-IPL-MGX treatment improve dry eye signs?

Participants were assigned to receive either three sessions of MBE-IPL-MGX treatment and home-based therapy (treatment group) or home-based therapy alone (control group).

The investigators will compare both groups to see if MBE-IPL-MGX treatment is superior to home-based therapy.

DETAILED DESCRIPTION:
MBE is a novel in-office treatment that works by exfoliating the eyelid margins to remove the accumulated biofilm debris, epithelial keratinization and capped meibomian glands, resulting in better meibum outflow . Different studies have shown that MBE improves DED symptoms [1,2], demodex blepharitis [1-4] and meibomian gland function [2,3,5] In addition, meta-analyses recommend combining IPL with meibomian gland expression (MGX) compared to IPL or MGX alone [6-8]. However, the investigators have not found any studies evaluating the benefits of MBE combined with IPL and MGX.

Consequently, the purpose of the current study is to evaluate whether MBE combined with IPL and MGX leads to an improvement of symptoms and signs in patients with DED due to MGD.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. DED diagnosis according to DEWS II meeting one of the following conditions: (2.1) ocular surface disease index (OSDI) score ≥ 13; (2.2) NIBUT < 10 seconds; and (2.3) ocular surface staining with > 5 or 9 corneal or conjunctival stains, respectively.
3. MGD diagnosis according to the international workshop on MGD meeting two of the following conditions: (3.1) irregularity of the eyelid margin or mucocutaneous junction; (3.2) vascularity of the eyelid margin; (3.3) plugged or capped Meibomian gland orifices; (3.4) Meibomian gland atrophy; or (3.5) decreased meibum quality and quantity

Exclusion Criteria:

1. Skin pathologies that prevent IPL treatment
2. All corneal disorders that affect diagnostic tests, such as: (2.1) active corneal infections; and (2.2) corneal dystrophies.
3. Active ocular allergy.
4. Pregnant or lactating women..
5. Patients who did not understand or comprehend the informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Ocular surface disease index (OSDI) questionnaire. | Change from Baseline OSDI at 2 months.
  Values from 0 (Better) to 100 (Worse)
Tear meniscus height (TMH) | Change from Baseline TMH at 2 months.
Tear meniscus area (TMA) | Change from Baseline TMA at 2 months.
Noninvasive tear film break-up time (NIBUT). | Change from Baseline NIBUT at 2 months.
Lipid Layer Grade (LLG) | Change from Baseline LLG at 2 months.
  Values from 0 (Better) to 4 (Worse)
Ciliary hyperemia | Change from Baseline Ciliary Hyperemia at 2 months.
  Values from 0 (Better) to 100 (Worse)
Conjunctival hyperemia | Change from Baseline Conjunctival Hyperemia at 2 months.
  Values from 0 (Better) to 100 (Worse)
Meibomian glands Loss area (LAMG) | Change from Baseline LAMG at 2 months.
  Values from 0 (Better) to 100 (Worse)
Meibomian gland secretions (MGS) | Change from Baseline MGS at 2 months.
  Values from 0 (Worse) to 45 (Better)
Meibomian gland Dysfunction Grade (MGD Grade) | Change from Baseline MGD grade at 2 months.
  Values from 0 (Better) to 4 (Worse)
Ocular surface staining (OSS). | Change from Baseline OSS at 2 months.
  Values from 0 (Better) to 4 (Worse)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Ballesteros Sánchez, Principal Investigator — University of Seville
Locations (1):
- Novovision ophthalmologic clinic, Murcia, Spain

REFERENCES:
- [Background] Murphy O, O'Dwyer V, Lloyd-McKernan A. The efficacy of tea tree face wash, 1, 2-Octanediol and microblepharoexfoliation in treating Demodex folliculorum blepharitis. Cont Lens Anterior Eye. 2018 Feb;41(1):77-82. doi: 10.1016/j.clae.2017.10.012. Epub 2017 Oct 23. PMID 29074306
- [Background] Mohammad-Rabei H, Arabi A, Shahraki T, Rezaee-Alam Z, Baradaran-Rafii A. Role of Blepharoexfoliation in Demodex Blepharitis: A Randomized Comparative Study. Cornea. 2023 Jan 1;42(1):44-51. doi: 10.1097/ICO.0000000000003046. Epub 2022 Apr 13. PMID 35439775
- [Background] Epstein IJ, Rosenberg E, Stuber R, Choi MB, Donnenfeld ED, Perry HD. Double-Masked and Unmasked Prospective Study of Terpinen-4-ol Lid Scrubs With Microblepharoexfoliation for the Treatment of Demodex Blepharitis. Cornea. 2020 Apr;39(4):408-416. doi: 10.1097/ICO.0000000000002243. PMID 31939919
- [Background] Siddireddy JS, Tan J, Vijay AK, Willcox MDP. The Effect of Microblepharon Exfoliation on Clinical Correlates of Contact Lens Discomfort. Optom Vis Sci. 2019 Mar;96(3):187-199. doi: 10.1097/OPX.0000000000001354. PMID 30801507
- [Background] Sambhi RS, Sambhi GDS, Mather R, Malvankar-Mehta MS. Intense pulsed light therapy with meibomian gland expression for dry eye disease. Can J Ophthalmol. 2020 Jun;55(3):189-198. doi: 10.1016/j.jcjo.2019.11.009. Epub 2020 Jan 13. PMID 31941589
- [Background] Leng X, Shi M, Liu X, Cui J, Sun H, Lu X. Intense pulsed light for meibomian gland dysfunction: a systematic review and meta-analysis. Graefes Arch Clin Exp Ophthalmol. 2021 Jan;259(1):1-10. doi: 10.1007/s00417-020-04834-1. Epub 2020 Jul 28. PMID 32725403
- [Background] Miao S, Yan R, Jia Y, Pan Z. Effect of Intense Pulsed Light Therapy in Dry Eye Disease Caused by Meibomian Gland Dysfunction: A Systematic Review and Meta-Analysis. Eye Contact Lens. 2022 Oct 1;48(10):424-429. doi: 10.1097/ICL.0000000000000934. Epub 2022 Sep 5. PMID 36044829

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/79/NCT05857579/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/79/NCT05857579/ICF_001.pdf